CLINICAL TRIAL: NCT02820480
Title: Design of an Affordable Gym for Post Stroke Rehabilitation
Acronym: RehabCares
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 823778
Record Dates: First submitted 2016-06-16; First posted 2016-07-01 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Stroke; Cerebral Palsy; Healthy
Keywords: stroke; rehabilitation; robotics; cerebral palsy; therapy
MeSH Terms: conditions — Stroke; Cerebral Palsy | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients/health professionals: Stroke AND cerebral palsy PATIENTS: greater than 18 years of age, who are more than 3 months post stroke, as well as health professionals who have considerable experience in stroke rehabilitation will be asked to evaluate the design of the Rehab in a Crate system. The aim is to survey stroke survivors and healthcare professionals on the design, ease of use, utility, and various features of, both existing and those yet-to-be-developed.
  Interventions: Device: Rehab in a Crate System

INTERVENTIONS:
Device: Rehab in a Crate System — The therapy gym is Rehab in a Crate with 4 stations for upper and lower limb assessment/therapy. Each station will allow adaptive game-based therapy.
  Note: The device is not being used at this moment for diagnostic or evaluation. Users will be asked to explore the device, try the systems, and provide feedback about use.

SUMMARY:
Rehab in a Crate is a therapy gym designed to be affordable, compact and easily transportable. The purpose of this particular study is to gain feedback on the initial design of the Rehab in a Crate system. This will be accomplished by using qualitative ethnographic research methods (i.e. human centered design) in the form of surveys that have been carefully designed by members of the research team. The eligibility criteria of this survey research reflects the intended user base of an eventual finished product, which is survivors of stroke and cerebral palsy across the globe. And while healthcare professionals are not the user base per se, their expertise and feedback should be instrumental in the design of future iterations of the Rehab in a Crate. Ease of use, utility, design, and various features, both existing and intended, will all be surveyed items.

DETAILED DESCRIPTION:
The investigators aim to survey stroke survivors and healthcare professionals on the design, ease of use, utility, and various features of, both existing and those yet-to-be-developed. This feedback will help to fine tune further development of this therapy gym, Rehab in a Crate, and move forward in the iteration process.

Note: The device is not being used at this moment for diagnostic or evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors who are more than 3 months post stroke and persons with cerebral palsy adults - have hemiplegia or diplegia
* Health professionals who have considerable experience in stroke rehabilitation.

Exclusion Criteria:

* Anyone who is not 18 years of age.
* More than mild spasticity in the upper of lower extremities.
* A cognitive score on the Montreal Cognitive Assessment that indicates that the participant is cognitively impaired.
* Motor impairment that precludes interaction with the Rehab in a Crate (e.g. unable to grip a handle).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Therapists and patients with neuro-rehab. Patients with neural injury
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Acceptability of Rehab system | 1 session, about 1.5 hours in length
  The ability to accept the product for use in rehab; An ethnographic survey/questionnaire will be administered to the subjects.

SECONDARY OUTCOMES:
Usability of Rehab System | 1 session, about 1.5 hours in length
  The ability to use the product for therapy as intended

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Johnson, PhD, Principal Investigator — Penn Medicine Rittenhouse
Locations (1):
- Penn Medicine Rittenhouse, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No